CLINICAL TRIAL: NCT01481779
Title: The Impact of LY2605541 Versus Insulin Glargine for Patients With Type 1 Diabetes Mellitus Treated With Preprandial Insulin Lispro: An Open-Label, Randomized, 78-Week Study - The IMAGINE 1 Study
Brief Title: A Study in Participants With Type 1 Diabetes Mellitus
Acronym: IMAGINE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12146; I2R-MC-BIAN (Other: Eli Lilly and Company); 2011-001261-40 (EudraCT Number)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; LY2605541; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2605541 + Insulin Lispro (Experimental): LY2605541 titrated based on blood glucose readings, administered by subcutaneous (SC) injection via pen device once daily at bedtime for 78 weeks in combination with Insulin Lispro. Insulin Lispro titrated based on blood glucose readings, administered by SC injection via pen device at meal times for 78 weeks.
  Interventions: Drug: LY2605541; Drug: Insulin Lispro
- Glargine + Insulin Lispro (Active Comparator): Glargine dose titrated based on blood glucose readings, administered by SC injection via pen device once daily at bedtime for 78 weeks in combination with Insulin Lispro. Insulin Lispro dose titrated based on blood glucose readings, administered by SC injection via pen device at meal times for 78 weeks.
  Interventions: Drug: Glargine; Drug: Insulin Lispro

INTERVENTIONS:
Drug: Glargine — Administered by SC injection via a pen device.
  Arms: Glargine + Insulin Lispro
Drug: LY2605541 — Administered by SC injection with a pen device.
  Arms: LY2605541 + Insulin Lispro
Drug: Insulin Lispro — Administered by SC injection with a pen device.
  Other Names: LY275585; Humalog

SUMMARY:
The purpose of this study is:

* To compare the blood sugar control of LY2605541 with insulin glargine after 78 weeks of treatment.
* To compare the rate of night-time low blood sugar episodes on LY2605541 with insulin glargine during 78 weeks of treatment.
* To compare the number of participants on LY2605541 reaching blood sugar targets without low blood sugar episodes at night to those taking insulin glargine after 78 weeks of treatment.
* To compare the rate of hypoglycemia episodes on LY2605541 with insulin glargine during 78 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have had diabetes mellitus for at least 1 year
* Have an hemoglobin A1c (HbA1c) value less than 12% according to the central laboratory at screening
* Have a body mass index (BMI) less than or equal to 35.0 kilograms per square meter (kg/m^2)
* Have been treated for at least 90 days prior to screening with the following:

  * Insulin detemir, insulin glargine, or human insulin isophane suspension (NPH) insulin in combination with premeal insulin,
  * Self-mixed or premixed insulin regimens with any basal and bolus insulin combination administered at least twice daily, or
  * Continuous SC insulin infusion therapy
* This inclusion criterion applies to female participants:

  * Are not breastfeeding
  * Test negative for pregnancy at screening and randomization based on serum pregnancy tests
  * Do not intend to become pregnant during the study
  * Have practiced a reliable method of birth control (for example, use of oral contraceptives or levonorgestrel, diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms with contraceptive foam, intrauterine devices, partner with vasectomy, or abstinence) for at least 6 weeks prior to screening
  * Agree to continue to use a reliable method of birth control during the study, as determined by the investigator (and for 2 weeks following the last dose of study drug)
* Capable of and willing and desirous to do the following: adhere to a multiple daily injection regimen, inject insulin with a prefilled pen and perform Self-Monitored Blood Glucose (SMBG) and record keeping as required by this protocol, as determined by the investigator. Caregiver may be responsible for all of the above.

Exclusion Criteria:

* Are using twice-daily insulin glargine having been inadequately controlled on once-daily dosed glargine prior to screening
* Have excessive insulin resistance defined as having received a total daily dose of insulin greater than 1.5 units per kilogram (units/kg) at the time of randomization
* Receiving any oral or injectable medication (other than metformin for treatment of polycystic ovarian disease) intended for the treatment of diabetes mellitus other than insulins in the 90 days prior to screening
* Lipid-lowering medications:

  * Are using niacin preparations as a lipid-lowering medication and/or bile acid sequestrants within 90 days prior to screening or are using lipid-lowering medication at a dose that has not been stable for greater than or equal to 90 days prior to screening
  * If a participant has not been on a stable dose of lipid-lowering medication for greater than or equal to 90 days prior to screening, the site should wait to screen the participant. If the results of the screening laboratory tests require a change to the participant's current lipid-lowering medication or initiation of lipid-lowering medication, it is acceptable to change the lipid-lowering medication for the participant and to have the participant return greater than or equal to 90 days later to complete some of the screening procedures again
* Have fasting hypertriglyceridemia (defined as greater than 4.5 millimoles per liter [mmol/L], greater than 400 milligrams per deciliter [mg/dL]) at screening, as determined by the central laboratory
* Have had more than 1 episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia as determined by the investigator) within 6 months prior to entry into the study
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control (hyperglycemia or diabetic ketoacidosis) in the past 6 months
* Cardiovascular: have cardiac disease with functional status that is New York Heart Association Class III or IV (per New York Heart Association Cardiac Disease Classification)
* Renal: Have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine greater than 2.5 mg/dL
* Hepatic: Have obvious clinical signs or symptoms of liver disease (excluding non-alcoholic fatty liver disease [NAFLD]), acute or chronic hepatitis, non-alcoholic steatohepatitis (NASH), or elevated liver enzyme measurements as indicated below:

  * Total bilirubin greater than or equal to 2 times the upper limit of normal (ULN) as defined by the central laboratory,
  * Alanine aminotransferase (ALT)/(serum glutamic pyruvic transaminase (SGPT) greater than 2.5 times ULN as defined by the central laboratory, or
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) greater than 2.5 times ULN as defined by the central laboratory.
* Malignancy: Have active or untreated malignancy, have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer) for less than 5 years, or are at an increased risk for developing cancer or a recurrence of cancer in the opinion of the investigator
* Allergy: Have known hypersensitivity or allergy to any of the study insulins or their excipients
* Hematologic: Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the HbA1c measurement
* Glucocorticoid therapy: Receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (excluding topical , intraocular, intranasal, and inhaled preparations) or have received such therapy within 8 weeks immediately before screening with the exception of replacement therapy for adrenal insufficiency
* Diagnosed clinically significant diabetic autonomic neuropathy, in the opinion of the investigator
* Have any other condition (including known drug or alcohol abuse or psychiatric disorder including eating disorder) that precludes the participant from following and completing the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (51):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntington Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Mateo, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- France (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bar-le-Duc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corbeil-Essonnes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Mandé
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vénissieux
- Germany (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eisenach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Falkensee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mayen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuwied
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pohlheim
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cagliari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lecce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perugia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ravenna
- Japan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara Jalisco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg

REFERENCES:
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287
- [Derived] Sanyal A, Cusi K, Hartman ML, Zhang S, Bastyr EJ 3rd, Bue-Valleskey JM, Chang AM, Haupt A, Jacober SJ, Konrad RJ, Zhang Q, Hoogwerf BJ. Cytokeratin-18 and enhanced liver fibrosis scores in type 1 and type 2 diabetes and effects of two different insulins. J Investig Med. 2018 Mar;66(3):661-668. doi: 10.1136/jim-2017-000609. Epub 2017 Nov 21. PMID 29167192
- [Derived] Orchard TJ, Cariou B, Connelly MA, Otvos JD, Zhang S, Antalis CJ, Ivanyi T, Hoogwerf BJ. The effects of basal insulin peglispro vs. insulin glargine on lipoprotein particles by NMR and liver fat content by MRI in patients with diabetes. Cardiovasc Diabetol. 2017 Jun 6;16(1):73. doi: 10.1186/s12933-017-0555-1. PMID 28587667
- [Derived] Cusi K, Sanyal AJ, Zhang S, Hartman ML, Bue-Valleskey JM, Hoogwerf BJ, Haupt A. Non-alcoholic fatty liver disease (NAFLD) prevalence and its metabolic associations in patients with type 1 diabetes and type 2 diabetes. Diabetes Obes Metab. 2017 Nov;19(11):1630-1634. doi: 10.1111/dom.12973. Epub 2017 Jun 22. PMID 28417532

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Started | 295 | 160
Received at Least 1 Dose of Study Drug | 294 | 159
Completed | 225 | 132
Not Completed | 70 | 28
Not completed — Adverse Event | 23 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 26 | 13
Not completed — Physician Decision | 13 | 4
Not completed — Sponsor Decision | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- LY2605541 + Insulin Lispro: LY2605541 titrated based on blood glucose readings, administered by SC injection via pen device once daily at bedtime for 78 weeks in combination with Insulin Lispro. Insulin Lispro titrated based on blood glucose readings, administered by SC injection via pen device at meal times for 78 weeks.
- Total: Total of all reporting groups
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro | Total
Number analyzed (Participants) | 295 | 160 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.68 (12.93) | 38.91 (14.10) | 39.41 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 73 | 230
  Male | 138 | 87 | 225
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 16 | 49
  Not Hispanic or Latino | 153 | 85 | 238
  Unknown or Not Reported | 109 | 59 | 168
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 9
  Asian | 63 | 31 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 221 | 125 | 346
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  France | 23 | 14 | 37
  United States | 85 | 45 | 130
  Mexico | 25 | 15 | 40
  Poland | 27 | 14 | 41
  Austria | 7 | 4 | 11
  Russia | 11 | 9 | 20
  Germany | 45 | 21 | 66
  Japan | 60 | 31 | 91
  Italy | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) at 26 Weeks
Description: HbA1c is a test that measures a participant's average blood glucose level over a 2- to 3-month timeframe. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM), adjusting for treatment, stratification factors (baseline low-density lipoprotein cholesterol [LDL-C] [<100 milligrams per deciliter (mg/dL) and ≥100 mg/dL] and country), visit, treatment-by-visit interaction, and baseline HbA1c as the fixed effects and participant as the random effect.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 287 | 153
percentage of HbA1c | 7.06 (0.04) | 7.43 (0.06)

2. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: HbA1c is a test that measures a participant's average blood glucose level over a 2- to 3-month timeframe. LS means were calculated using MMRM, adjusting for treatment, stratification factors (baseline LDL-C [<100 mg/dL and ≥100 mg/dL] and country), visit, treatment-by-visit interaction, and baseline HbA1c as the fixed effects.
Time Frame: 52 weeks and 78 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 287 | 153
percentage of HbA1c
  Week 52 | 7.30 (0.05) | 7.55 (0.06)
  Week 78 | 7.43 (0.05) | 7.70 (0.07)

3. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: as for outcome 2
Time Frame: Baseline, 26 weeks, 52 weeks, 78 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 287 | 153
percentage of HbA1c
  Week 26 | -0.69 (0.04) | -0.33 (0.06)
  Week 56 | -0.46 (0.05) | -0.21 (0.06)
  Week 78 | -0.33 (0.05) | -0.05 (0.07)

4. Secondary Outcome: Percentage of Participants With Hemoglobin A1c (HbA1c) Less Than 7.0% or Less Than or Equal to 6.5% Using Last Observation Carried Forward (LOCF)
Description: HbA1c is a test that measures a participant's average blood glucose level over a 2- to 3-month timeframe. The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, then multiplying by 100.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data. Missing endpoints were imputed with the LOCF method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 287 | 153
percentage of participants
  HbA1c ≤6.5%, Week 26 | 28.6 | 13.7
  HbA1c ≤6.5%, Week 52 | 23.3 | 13.1
  HbA1c ≤6.5%, Week 78 | 20.2 | 13.1
  HbA1c <7.0%, Week 26 | 44.9 | 27.5
  HbA1c <7.0%, Week 52 | 37.3 | 28.1
  HbA1c <7.0%, Week 78 | 34.5 | 22.9

5. Secondary Outcome: Proportion of Participants With Hemoglobin A1c (HbA1c) Less Than 7.0% Without Nocturnal Hypoglycemia
Description: Hypoglycemic episodes are defined as an event that is associated with reported signs and symptoms of hypoglycemia and/or a documented blood glucose concentration of ≤70 mg/dL (3.9 millimoles per liter [mmol/L]). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. The percentage of participants was calculated by dividing the number of participants with HbA1c <7.0% without nocturnal hypoglycemia by the total number of participants analyzed, then multiplying by 100.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable data. Missing endpoints were imputed with the LOCF method.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 287 | 153
percentage of participants
  Week 26 | 3.8 | 2.0
  Week 52 | 2.1 | 0.7
  Week 78 | 1.0 | 0.0

6. Secondary Outcome: Total Hypoglycemia Rates (Adjusted by 30 Days)
Description: Hypoglycemic episodes are defined as events that are associated with reported signs and symptoms of hypoglycemia and/or documented blood glucose (BG) concentrations of ≤70 mg/dL (3.9 mmol/L). Group mean rates of total hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models (number of episodes = treatment + baseline total hypoglycemia rate, with log [exposure in days/30] as an offset variable). Group mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks and Baseline through 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable data at both baseline and post-baseline.
Measure: Mean (Standard Error); unit: episodes/participant/30 days
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 293 | 159
episodes/participant/30 days
  Baseline-Week 26 | 16.01 (0.44) | 12.43 (0.55)
  Baseline-Week 52 | 14.84 (0.42) | 11.75 (0.55)
  Baseline-Week 78 | 14.33 (0.42) | 11.43 (0.55)

7. Secondary Outcome: Percentage of Participants With Total Hypoglycemia Events
Description: Hypoglycemic events are defined as events that are associated with reported signs and symptoms of hypoglycemia and/or documented BG concentrations of ≤70 mg/dL (3.9 mmol/L). The percentage of participants was calculated by dividing the number of participants with hypoglycemic episodes by the total number of participants analyzed, then multiplying by 100.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks and Baseline through 78 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 294 | 159
percentage of participants
  Baseline-Week 26 | 99.0 | 96.9
  Baseline-Week 52 | 99.0 | 96.9
  Baseline-Week 78 | 99.0 | 96.9

8. Secondary Outcome: Nocturnal Hypoglycemia Rates (Adjusted by 30 Days)
Description: Hypoglycemic episodes are defined as events that are associated with reported signs and symptoms of hypoglycemia and/or a documented BG concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. Group mean rates of nocturnal hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models (number of episodes = treatment + baseline nocturnal hypoglycemia rate, with log [exposure in days/30] as an offset variable). Group mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks and Baseline through 78 weeks
Population: as for outcome 6
Measure: Mean (Standard Error); unit: episodes/participant/30 days
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 293 | 159
episodes/participant/30 days
  Baseline-Week 26 | 1.69 (0.12) | 2.66 (0.19)
  Baseline-Week 52 | 1.63 (0.11) | 2.45 (0.19)
  Baseline-Week 78 | 1.58 (0.11) | 2.28 (0.17)

9. Secondary Outcome: Percentage of Participants With Nocturnal Hypoglycemic Events
Description: Hypoglycemic episodes are defined as an event that is associated with reported signs and symptoms of hypoglycemia and/or a BG concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. The percentage of participants was calculated by dividing the number of participants with nocturnal hypoglycemic episodes by the total number of participants analyzed, then multiplying by 100.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks and Baseline through 78 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 294 | 159
percentage of participants
  Baseline-Week 26 | 87.4 | 90.6
  Baseline-Week 52 | 91.5 | 91.8
  Baseline-Week 78 | 93.5 | 92.5

10. Secondary Outcome: Fasting Serum Glucose (FSG) by Laboratory Measurement
Description: LS means were calculated using MMRM, adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], baseline LDL-C level [<100 mg/dL and ≥100 mg/dL], and country), visit, treatment-by-visit interaction, and corresponding baseline dependent variable as the fixed effects, and participants as the random effect.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable FSG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 285 | 152
mg/dL
  Week 26 | 138.22 (3.80) | 160.35 (5.06)
  Week 52 | 146.55 (4.42) | 164.28 (5.72)
  Week 78 | 144.64 (4.53) | 164.78 (5.81)

11. Secondary Outcome: Fasting Blood Glucose (FBG) Intra-participant Variability
Description: FBG was measured by self-monitored blood glucose (SMBG). Between-day glucose variability is measured by the standard deviation of FBG. LS means were calculated using MMRM, adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], baseline LDL-C level [<100 mg/dL and ≥100 mg/dL], and country), visit, treatment-by-visit interaction, and corresponding baseline dependent variable as the fixed effects, and participants as the random effect.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable FBG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 282 | 153
mg/dL
  Week 26 | 52.49 (1.79) | 59.25 (2.43)
  Week 52 | 53.44 (1.85) | 58.15 (2.43)
  Week 78 | 54.87 (2.20) | 60.66 (2.79)

12. Secondary Outcome: 0300-hour Blood Glucose (BG) to Fasting Blood (FBG) Glucose Excursion
Description: Results of a 0300-hour to pre-morning meal (FBG) excursion are presented (only SMBG profiles with both 0300 hours and the next day pre-morning measurements are included for the calculation of such excursion). LS means were calculated using MMRM, adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], baseline LDL-C level [<100 mg/dL and ≥100 mg/dL], and country), visit, treatment-by-visit interaction, and corresponding baseline dependent variable as the fixed effects and participants as the random effect.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable SMBG data at baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 209 | 112
mg/dL
  Week 26 | -9.92 (6.24) | -14.08 (8.75)
  Week 52 | -6.15 (6.91) | -9.02 (9.58)
  Week 78 | -10.82 (8.25) | -28.94 (10.50)

13. Secondary Outcome: 9 Point Self-monitored Blood Glucose (SMBG)
Description: 9-point SMBG profiles were obtained over 2 days within the week prior to Weeks 0, 4, 12, 26, 39, 52, 65, and 78. SMBG measurements were taken at 9 time points: pre-morning meal, 2 hours post-morning meal, pre-midday meal, 2 hours post-midday meal, pre-evening meal, 2 hours post-evening meal, bedtime, at approximately 0300 hours, and the pre-morning meal the next day. LS means were calculated using MMRM, adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], baseline LDL-C level [<100 mg/dL and ≥100 mg/dL], and country), visit, treatment-by-visit interaction, and corresponding baseline dependent variable as the fixed effects and participants as the random effect.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable SMBG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 271 | 143
mg/dL
  Pre-morning meal, Week 26 | 158.58 (3.82) | 144.40 (5.20)
  Pre-morning meal, Week 52 | 160.89 (4.13) | 152.55 (5.38)
  Pre-morning meal, Week 78 | 163.09 (4.66) | 153.38 (5.99)
  2 hours post-morning meal, Week 26: number analyzed (Participants) | 245 | 125
  2 hours post-morning meal, Week 26 | 172.39 (4.59) | 165.53 (6.44)
  2 hours post-morning meal, Week 52: number analyzed (Participants) | 245 | 125
  2 hours post-morning meal, Week 52 | 176.32 (5.61) | 168.38 (7.47)
  2 hours post-morning meal, Week 78: number analyzed (Participants) | 245 | 125
  2 hours post-morning meal, Week 78 | 183.64 (6.23) | 190.54 (7.91)
  Pre-midday meal, Week 26: number analyzed (Participants) | 264 | 140
  Pre-midday meal, Week 26 | 136.21 (3.92) | 153.12 (5.33)
  Pre-midday meal, Week 52: number analyzed (Participants) | 264 | 140
  Pre-midday meal, Week 52 | 142.82 (4.27) | 149.78 (5.66)
  Pre-midday meal, Week 78: number analyzed (Participants) | 264 | 140
  Pre-midday meal, Week 78 | 150.83 (4.90) | 154.56 (6.33)
  2 hours post-midday meal, Week 26: number analyzed (Participants) | 244 | 122
  2 hours post-midday meal, Week 26 | 157.17 (4.78) | 164.75 (6.69)
  2 hours post-midday meal, Week 52: number analyzed (Participants) | 244 | 122
  2 hours post-midday meal, Week 52 | 159.59 (5.11) | 168.83 (6.94)
  2 hours post-midday meal, Week 78: number analyzed (Participants) | 244 | 122
  2 hours post-midday meal, Week 78 | 154.46 (5.76) | 175.52 (7.51)
  Pre-evening meal, Week 26: number analyzed (Participants) | 266 | 143
  Pre-evening meal, Week 26 | 153.20 (4.29) | 168.08 (5.75)
  Pre-evening meal, Week 52: number analyzed (Participants) | 266 | 143
  Pre-evening meal, Week 52 | 153.01 (5.17) | 183.18 (6.81)
  Pre-evening meal, Week 78: number analyzed (Participants) | 266 | 143
  Pre-evening meal, Week 78 | 149.89 (4.92) | 174.50 (6.17)
  2 hours post-evening meal, Week 26: number analyzed (Participants) | 232 | 126
  2 hours post-evening meal, Week 26 | 149.74 (5.17) | 191.99 (7.20)
  2 hours post-evening meal, Week 52: number analyzed (Participants) | 232 | 126
  2 hours post-evening meal, Week 52 | 157.81 (6.79) | 198.10 (9.06)
  2 hours post-evening meal, Week 78: number analyzed (Participants) | 232 | 126
  2 hours post-evening meal, Week 78 | 163.27 (6.07) | 189.43 (7.75)
  Bedtime, Week 26: number analyzed (Participants) | 250 | 137
  Bedtime, Week 26 | 151.66 (4.15) | 176.17 (5.63)
  Bedtime, Week 52: number analyzed (Participants) | 250 | 137
  Bedtime, Week 52 | 167.35 (5.33) | 182.08 (7.11)
  Bedtime, Week 78: number analyzed (Participants) | 250 | 137
  Bedtime, Week 78 | 165.63 (5.37) | 185.45 (6.74)
  0300 hours, Week 26: number analyzed (Participants) | 219 | 116
  0300 hours, Week 26 | 159.73 (5.30) | 163.18 (7.50)
  0300 hours, Week 52: number analyzed (Participants) | 219 | 116
  0300 hours, Week 52 | 157.52 (6.06) | 148.26 (8.36)
  0300 hours, Week 78: number analyzed (Participants) | 219 | 116
  0300 hours, Week 78 | 165.82 (7.19) | 170.35 (9.02)
  Pre-morning meal next day, Week 26: number analyzed (Participants) | 260 | 138
  Pre-morning meal next day, Week 26 | 149.94 (3.74) | 143.89 (5.10)
  Pre-morning meal next day, Week 52: number analyzed (Participants) | 260 | 138
  Pre-morning meal next day, Week 52 | 155.79 (4.24) | 145.55 (5.59)
  Pre-morning meal next day, Week 78: number analyzed (Participants) | 260 | 138
  Pre-morning meal next day, Week 78 | 156.87 (4.80) | 152.63 (6.11)

14. Secondary Outcome: Change From Baseline in Body Weight
Description: as for outcome 10
Time Frame: Baseline and 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable body weight data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 287 | 154
kilograms (kg)
  Week 26 | -1.17 (0.20) | 0.71 (0.27)
  Week 52 | -1.22 (0.25) | 1.00 (0.33)
  Week 78 | -0.93 (0.28) | 1.04 (0.37)

15. Secondary Outcome: Basal, Bolus, and Total Insulin Dose
Description: Basal insulin dose, short-acting bolus insulin dose (each meal and overall), and total insulin dose were calculated based on the dose during the last 7 days prior to the post-treatment visit or last 3 days prior to the randomization visit. LS means were calculated using MMRM, adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], baseline LDL-C level [<100 mg/dL and ≥100 mg/dL], and country), visit, treatment-by-visit interaction, and corresponding baseline dependent variable as the fixed effects and participants as the random effect.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: units/kg/day
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 282 | 156
units/kg/day
  Basal Insulin, Week 26: number analyzed (Participants) | 239 | 127
  Basal Insulin, Week 26 | 0.40 (0.01) | 0.34 (0.01)
  Basal Insulin, Week 52: number analyzed (Participants) | 239 | 127
  Basal Insulin, Week 52 | 0.40 (0.01) | 0.34 (0.01)
  Basal Insulin, Week 78: number analyzed (Participants) | 239 | 127
  Basal Insulin, Week 78 | 0.41 (0.01) | 0.35 (0.01)
  Bolus Insulin, Week 26: number analyzed (Participants) | 280 | 153
  Bolus Insulin, Week 26 | 0.37 (0.01) | 0.46 (0.02)
  Bolus Insulin, Week 52: number analyzed (Participants) | 280 | 153
  Bolus Insulin, Week 52 | 0.38 (0.01) | 0.47 (0.02)
  Bolus Insulin, Week 78: number analyzed (Participants) | 280 | 153
  Bolus Insulin, Week 78 | 0.37 (0.02) | 0.48 (0.02)
  Total Insulin, Week 26 | 0.73 (0.02) | 0.78 (0.02)
  Total Insulin, Week 52 | 0.74 (0.02) | 0.79 (0.03)
  Total Insulin, Week 78 | 0.75 (0.02) | 0.80 (0.03)

16. Secondary Outcome: Lipid Profile
Description: Concentrations of cholesterol, high-density lipoprotein cholesterol (HDL-C), LDL-C, and triglycerides are summarized. LS means were calculated using MMRM, adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, LDL-C [<100 mg/dL and ≥100 mg/dL] except for the LDL-C outcome variable), visit, treatment, treatment-by-visit interaction, and baseline value of corresponding lipid outcome variable.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable lipid data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 288 | 152
mg/dL
  Cholesterol, Week 26 | 191.86 (1.63) | 187.93 (2.19)
  Cholesterol, Week 52 | 190.72 (1.59) | 188.65 (2.10)
  Cholesterol, Week 78 | 191.78 (1.86) | 190.06 (2.39)
  HDL-C, Week 26 | 61.87 (0.59) | 62.75 (0.80)
  HDL-C, Week 52 | 61.01 (0.56) | 61.46 (0.74)
  HDL-C, Week 78 | 60.77 (0.66) | 61.97 (0.85)
  LDL-C, Week 26 | 108.85 (1.33) | 108.31 (1.79)
  LDL-C, Week 52 | 109.40 (1.39) | 109.74 (1.84)
  LDL-C, Week 78 | 109.62 (1.62) | 110.35 (2.09)
  Triglycerides, Week 26 | 109.64 (3.89) | 85.35 (5.24)
  Triglycerides, Week 52 | 105.17 (3.64) | 87.94 (4.80)
  Triglycerides, Week 78 | 110.80 (4.78) | 88.96 (6.14)

17. Secondary Outcome: Percentage of Participants With Change in Anti-LY2605541 Antibodies
Description: The percentage of participants with a treatment-emergent anti-LY2605541 antibody response (TEAR) is summarized. TEAR is defined as change from baseline to post-baseline in the anti-LY2605541 antibody level either from undetectable to detectable or from detectable to the value with at least 130% relative increase from baseline.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks and Baseline through 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable anti-LY2605541 antibody data at baseline and post-baseline. Missing endpoints were imputed with the LOCF method.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 288 | 153
percentage of participants
  Week 26: number analyzed (Participants) | 288 | 152
  Week 26 | 30.6 | 15.8
  Week 52: number analyzed (Participants) | 288 | 152
  Week 52 | 29.9 | 17.1
  Week 78 | 26.4 | 13.1

18. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ)
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, and Insulin Delivery Device. Data presented are the transformed overall score on a scale of 0-100, where higher scores indicate better treatment satisfaction. LS means were calculated using an analysis of covariance (ANCOVA) model with treatment and stratification (baseline HbA1c [≤8.5% or >8.5%] and country) as fixed effects and baseline value of the dependent variable as a covariate.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable ITSQ data at both baseline and post-baseline. Missing endpoints were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 273 | 149
units on a scale | 72.43 (0.69) | 73.91 (0.94)

19. Secondary Outcome: Low Blood Sugar Survey (LBSS)
Description: LBSS (also referenced as Hypoglycemia Fear Survey - II [HFS-II]) is a 33-item questionnaire that measures 1) behaviors to avoid hypoglycemia and its negative consequences (15 items) and 2) worries about hypoglycemia and its negative consequences (18 items). Responses are made on a 5-point Likert scale where 0 = Never and 4 = Always. Total score is the sum of all items (range 0-132). Higher total scores reflect greater fear of hypoglycemia. LS means were calculated using MMRM, adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%] and country), visit, treatment-by-visit interaction , and corresponding baseline dependent variable as the fixed effects and participants as the random effect.
Time Frame: 26 weeks and 52 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable LBSS data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 287 | 151
units on a scale
  Week 26 | 28.09 (0.70) | 27.09 (0.95)
  Week 52 | 27.76 (0.77) | 27.00 (1.01)
  Week 78 | 27.68 (0.91) | 27.14 (1.18)

20. Secondary Outcome: European Quality of Life-5 Dimension (EQ-5D)
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) using a 3-level scale of 1-3 (no problem, some problems, and extreme problems). These combinations of attributes are converted into a weighted health-state Index Score according to the United States population-based algorithm. Scores range from -0.11 to 1.0, where a score of 1.0 indicates perfect health. LS means were calculated using ANCOVA, adjusting for treatment and stratification factors (baseline HbA1c [≤8.5% or >8.5%] and country) as fixed effects and baseline EQ-5D score as a covariate.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable EQ-5D data at both baseline and post-baseline. Missing endpoints were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 277 | 150
units on a scale | 0.92 (0.01) | 0.91 (0.01)

21. Secondary Outcome: Rapid Assessment of Physical Activity (RAPA)
Description: The RAPA questionnaire assesses the level and intensity of physical activity of adult participants. It contains 2 subscales: RAPA 1 (Aerobic) and RAPA 2 (Strength and Flexibility). RAPA 1 contains 7 questions regarding the participant's amount and intensity of physical activity, allowing each participant's aerobic activity level to be categorized as sedentary, underactive, light activities, light activity, regular underactive, or active. RAPA 2 contains 2 questions regarding participants' physical activities that increase strength and improve flexibility. Each participant's strength and flexibility activity level is then categorized as neither strength nor flexibility (flex) activity, either strength or flex (not both), both strength and flex activity. The percentage of participants in each RAPA 1/2 category is presented and was calculated by dividing the number of participants in each RAPA 1/2 category by the total number of participants analyzed, then multiplying by 100.
Time Frame: 26 weeks and 78 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable RAPA data. Missing endpoints were imputed with the LOCF method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Number analyzed (Participants) | 98 | 57
percentage of participants
  RAPA 1, Sedentary, Week 26 | 1.0 | 0.0
  RAPA 1, Sedentary, Week 78: number analyzed (Participants) | 80 | 51
  RAPA 1, Sedentary, Week 78 | 1.3 | 0.0
  RAPA 1, Underactive, Week 26 | 3.1 | 3.5
  RAPA 1, Underactive, Week 78: number analyzed (Participants) | 80 | 51
  RAPA 1, Underactive, Week 78 | 3.8 | 2.0
  RAPA 1, Light activity, Week 26 | 13.3 | 10.5
  RAPA 1, Light activity, Week 78: number analyzed (Participants) | 80 | 51
  RAPA 1, Light activity, Week 78 | 7.5 | 13.7
  RAPA 1, Regular underactive, Week 26 | 24.5 | 29.8
  RAPA 1, Regular underactive, Week 78: number analyzed (Participants) | 80 | 51
  RAPA 1, Regular underactive, Week 78 | 31.3 | 29.4
  RAPA 1, Active, Week 26 | 58.2 | 56.1
  RAPA 1, Active, Week 78: number analyzed (Participants) | 80 | 51
  RAPA 1, Active, Week 78 | 56.3 | 54.9
  RAPA 2, Neither strength/flex, Week 26 | 35.7 | 43.9
  RAPA 2, Neither strength/flex, Week 78: number analyzed (Participants) | 81 | 51
  RAPA 2, Neither strength/flex, Week 78 | 37.0 | 47.1
  RAPA 2, Either strength/flex, Week 26 | 30.6 | 35.1
  RAPA 2, Either strength/flex, Week 78: number analyzed (Participants) | 81 | 51
  RAPA 2, Either strength/flex, Week 78 | 33.3 | 29.4
  RAPA 2, Both strength/flex, Week 26 | 33.7 | 21.1
  RAPA 2, Both strength/flex, Week 78: number analyzed (Participants) | 81 | 51
  RAPA 2, Both strength/flex, Week 78 | 29.6 | 23.5

ADVERSE EVENTS:
Groups:
- LY2605541 + Insulin Lispro: LY2605541 titrated based on blood glucose readings, administered by subcutaneous (SC) injection via pen device once daily at bedtime for 78 weeks in combination with Insulin Lispro. Insulin Lispro titrated based on blood glucose readings, administered subcutaneously via pen device at meal times for 78 weeks.
Arm/Group | LY2605541 + Insulin Lispro | Glargine + Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 67/294 | 25/159
Other Adverse Events (participants affected / at risk) | 256/294 | 112/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2605541 + Insulin Lispro (N=294) | Glargine + Insulin Lispro (N=159)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (4)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Faeces pale (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (3) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (4) | 1 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 45 (73) | 13 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/157 (1) | 0/73 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/157 (5) | 0/73 (0)
Complicated migraine (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (3) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (3) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1/157 (2) | 0/73 (0)
Menorrhagia (Reproductive system and breast disorders) | 1/157 (2) | 0/73 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1/157 (2) | 0/73 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1/157 (1) | 0/73 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 + Insulin Lispro (N=294) | Glargine + Insulin Lispro (N=159)
Diarrhoea (Gastrointestinal disorders) | 13 (15) | 3 (3)
Bronchitis (Infections and infestations) | 11 (12) | 4 (4)
Cystitis (Infections and infestations) | 9 (10) | 3 (3)
Gastroenteritis (Infections and infestations) | 11 (11) | 8 (9)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 5 (6)
Influenza (Infections and infestations) | 25 (32) | 14 (14)
Nasopharyngitis (Infections and infestations) | 92 (152) | 38 (61)
Pharyngitis (Infections and infestations) | 13 (19) | 7 (9)
Upper respiratory tract infection (Infections and infestations) | 13 (22) | 12 (17)
Urinary tract infection (Infections and infestations) | 15 (17) | 8 (14)
Alanine aminotransferase increased (Investigations) | 12 (20) | 1 (1)
Weight increased (Investigations) | 4 (4) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 7 (7)
Headache (Nervous system disorders) | 18 (27) | 10 (13)
Depression (Psychiatric disorders) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 5 (6)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 17 (24) | 1 (1)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 45 (66) | 0 (0)
Hypertension (Vascular disorders) | 10 (10) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days